CLINICAL TRIAL: NCT04243252
Title: Healthy Pantry Program Intervention Evaluation (HAPPIE)
Brief Title: A Trial of Traffic Light Labeling With Behavioral Nudges and a Healthy Recipe Database to Increase Selection of Healthier Foods in Client-choice Food Pantries
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID pandemic
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Greater Boston Food Bank (Unknown)
Responsible Party: Principal Investigator, Anne N. Thorndike, MD, MPH, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019P003211
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Food Selection
Keywords: food insecurity
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Food Pantries (Experimental): Food pantries will complete online training to help them rank foods by nutritional value and promote those foods to pantry clients; the effect on pantries and their clients will be measured.
  Interventions: Behavioral: Healthy Pantry Program
- Control Food Pantries (Active Comparator): Food pantries will continue to operate as usual during the study period; the effect on pantries and their clients will be measured.
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Behavioral: Healthy Pantry Program — Food pantries will receive the Healthy Pantry Program online training, which will be completed by at least one pantry staff member and teaches pantry staff a novel traffic-light nutrition labeling system, a multilingual healthy recipe database, and how to use those and other behavioral economic strategies to implement simple interventions in the food pantry to promote client selection of healthier options. Onsite support by a registered dietitian is included.
  Arms: Intervention Food Pantries
Other: Waitlist Control — Normal food pantry use for duration of the 9-month study period. Control pantries will have access to the Healthy Pantry Program after study is completed.
  Arms: Control Food Pantries

SUMMARY:
This study is a pilot evaluation of the Healthy Pantry Program, a new behavioral economics-based training that allows pantry staff to learn how to implement nudges integrating traffic-light nutrition labeling and a healthy recipe database in the pantry environment. The hypothesis is that participation the Healthy Pantry Program will lead to increases in pantry purchases of healthy foods.

DETAILED DESCRIPTION:
Food insecurity affects more than one in 10 Americans and is associated with poor nutrition and adverse health outcomes, including diabetes, hypertension, and mental health issues. Many food-insecure individuals use food pantries, which provide charitable food, to supplement household food needs. The emergence of client-choice food pantries, where individuals can select the foods they take home, provides a novel opportunity to intervene on the diets of food pantry clients.

This study evaluates the Healthy Pantry Program (HPP) in a sample of 10 food pantries in the greater Boston area. Pantries will be matched on baseline characteristics and randomized 1:1 into participation in HPP (intervention) or wait list (control). Outcomes data will be collected at the pantry and client level. The aims of the study are as follows:

Aim 1: To evaluate whether HPP is associated with increased healthy food purchases from the food bank by intervention food pantries compared to control food pantries.

Aim 2: To evaluate whether HPP is associated with increases in the availability of healthy food in intervention food pantries compared to control food pantries.

Aim 3: To evaluate whether HPP is associated with an increase in healthy food selection and dietary intake by clients of intervention food pantries compared to clients of control food pantries, using a cross-sectional sample of 400 food pantry clients at baseline and 400 food pantry clients at 6-month follow up.

ELIGIBILITY:
Pantry Inclusion Criteria:

* maximum client-choice (clients can choose all items that they take from pantry)
* operate at least once weekly
* affiliated with the Greater Boston Food Bank

Pantry Exclusion Criteria:

* not affiliated with the Greater Boston Food Bank
* operating less than once weekly
* not a maximum client-choice food pantry
* >1 hr drive from Boston
* <50 clients on average per open day

Client Inclusion Criteria (for cross-sectional surveys at baseline and 6-month follow up):

* ≥18 years old
* pantry client
* speaks English or Spanish

Client Exclusion Criteria:

* <18 years old
* does not speak English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Monthly change in proportion of green-labeled foods purchased by food pantries from the food bank | Collected from the electronic ordering system at baseline and prospectively each month for 9 months
  Monthly change from baseline values of healthier foods purchased by pantries from the food bank in the proportion of green-labeled foods.
Monthly change in the Healthy Purchasing Score of foods purchased by food pantries from the food bank | Collected from the electronic ordering system at baseline and prospectively each month for 9 months
  Monthly change from baseline values of healthier foods purchased by pantries from the food bank in a weighted Healthy Purchasing Score that includes all foods (range: 0-1, higher scores represent healthier selection)

SECONDARY OUTCOMES:
Change in food availability at food pantries | Assessed at baseline and 6 months
  Change from baseline in food availability score using the Healthy Food Pantry Assessment Tool (range: 0-45, higher scores represent greater food availability)
Change in healthier food selection by pantry clients | Assessed at baseline and 6 months
  Change from baseline in pantry basket inventories of pantry clients measured by the proportion of green-labeled foods for each basket
Change in healthier food selection by pantry clients | Assessed at baseline and 6 months
  Change from baseline in pantry basket inventories of pantry clients measured by Healthy Purchasing Score for each basket (range: 0-1, higher scores represent healthier selection)
Change in self-reported fruit and vegetable intake of pantry clients | Assessed at baseline and 6 months
  Change from baseline fruit and vegetable intake in cup equivalents measured by the Dietary Screener from the California Health Information Survey 2005

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No